CLINICAL TRIAL: NCT07320703
Title: "Breathlessness Diagnostics in a Box" (BiaB) for Primary Care. A Multi-country Quality Improvement Project Using a Randomized Stepped-wedge Design
Acronym: BiaB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Practitioners Research Institute (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GPRI-2024-001; EUPAS1000000217 (Other: EU PAS Register)
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breathlessness; Cardiovascular; Pulmonary; Mental Disease
Keywords: breathlessness; diagnostics; cardiovascular disease; pulmonary disease; mental disease; cardiopulmonary risk
MeSH Terms: conditions — Dyspnea; Mental Disorders; Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Intervention Model Description: A prospective stepped-wedge study design will be used for this study. In every country, participating sites will be assigned to one of the five sequences (3 sites per sequence) for timing of the intervention start. Each sequence starts with a usual care period (6 weeks or a multiple of 6) which will be followed by a transition period of 4 weeks prior to the BiaB intervention period (6 weeks or a multiple of 6). During the transition period the healthcare professionals (HCPs) at the site will be instructed about the start date of the BiaB intervention and they will receive training for the use of BiaB. The study duration for sites is 40 weeks in total. The maximum study duration for patients is one visit followed by a maximum of 4 quarterly questionnaires (1 year).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Patients are managed according to usual care for the assessment of breathlessness in general practice, without use of the Breathlessness diagnostics in a Box (BiaB) tool. Clinical assessments, diagnostic procedures, and follow-up are performed as part of routine practice. Data collected during this period are used as control data for comparison with the intervention period.
- BiaB Intervention (Experimental): Patients are managed using the Breathlessness diagnostics in a Box (BiaB) tool as part of routine clinical care. The BiaB intervention supports general practitioners in the diagnostic assessment of patients presenting with breathlessness. No study-mandated therapeutic interventions are applied. Outcomes during the intervention period are compared with those from the usual care period.
  Interventions: Diagnostic Test: Breathlessness diagnostics in a Box (BiaB)

INTERVENTIONS:
Diagnostic Test: Breathlessness diagnostics in a Box (BiaB) — The Breathlessness diagnostics in a Box (BiaB) is a diagnostic support tool used in general practice to assist healthcare professionals in the assessment of patients presenting with breathlessness as part of routine clinical care.
  Arms: BiaB Intervention

SUMMARY:
This prospective stepped-wedge study evaluates whether use of the Breathlessness diagnostics in a Box (BiaB) tool shortens the time to diagnosis in patients presenting with breathlessness, compared with usual care. The study is conducted in general practice settings in the Netherlands, Spain, and Portugal. Participating sites start with a usual care period and transition sequentially to the BiaB intervention period. Data are collected during routine clinical visits, from electronic medical records, and through questionnaires completed by patients and healthcare professionals.

DETAILED DESCRIPTION:
This is a prospective interventional study using a stepped-wedge cluster design with a usual care period followed by an intervention period. Participating general practice sites are assigned to one of five predefined sequences determining the timing of transition from usual care to the BiaB intervention. All sites start in the usual care phase and sequentially transition to the intervention phase according to the study schedule.

The primary objective of the study is to assess whether use of BiaB shortens the time to diagnosis in patients presenting with breathlessness, compared with usual care without BiaB. Secondary objectives include evaluating whether BiaB increases the number of new diagnoses of chronic obstructive pulmonary disease (COPD) and cardiovascular disease (CVD), and assessing the usability and efficiency of the BiaB tool.

The study is conducted in general practice settings in the Netherlands, Spain, and Portugal, with a total of 45 sites. Each site participates for a total duration of 40 weeks. Patients attend a single study visit and may complete up to four quarterly questionnaires over a maximum follow-up of one year. Data are collected during routine clinical care, from electronic medical records, and via questionnaires completed by patients and healthcare professionals. Data from the usual care period, and where available retrospective data, are used as control data for comparison with the intervention period.

ELIGIBILITY:
The study aims to capture the real-world heterogeneity in primary care practices and patients. Therefore, inclusion and exclusion criteria are limited.

Inclusion criteria

* Patient must be at least 18 years old at the time of signing the informed consent.
* Patients that present with undiagnosed dyspnea (breathlessness); or Patients who have existing diseases that could cause breathlessness, but have residual or increasing breathlessness that could be caused by other not yet detected diseases. Or HCP has doubts or requires additional tests to confirm diagnosis or to suspect new, parallel, diagnoses. For example, breathlessness in patients assessed within the framework of Cardiovascular Risk Management or for COPD monitoring

Exclusion criteria

1. Acute worsening of previous diagnosed chronic disease where there is no suspicion of comorbidities (for example when a patient with clear COPD diagnosis has an exacerbation where typically the HCP will not perform additional tests).
2. Inability to understand and sign the written consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of the cause of breathlessness | From first presentation or consultation for breathlessness up to the date of diagnosis, assessed during the study period (up to 40 weeks per site).
  Number of days between the first presentation or consultation for breathlessness and the date of diagnosis of the underlying cause of breathlessness, comparing periods of usual care and periods with use of the Breathlessness diagnostics in a Box (BiaB) intervention.

SECONDARY OUTCOMES:
Number of new diagnoses of COPD and cardiovascular disease | Assessed during the study period (up to 40 weeks per site).
  Number of newly diagnosed cases of chronic obstructive pulmonary disease (COPD) and cardiovascular disease (CVD) identified during periods of usual care compared with periods with use of the Breathlessness diagnostics in a Box (BiaB) intervention.
Usability and efficiency of the BiaB tool | During the intervention period, with follow-up questionnaires completed up to 12 months after the index visit.
  Usability and efficiency of the Breathlessness diagnostics in a Box (BiaB) tool as assessed by questionnaires completed by healthcare professionals and patients during the intervention period.

CONTACTS AND LOCATIONS:
Locations (3):
- 15 primary care sites across the Netherlands, Groningen, Netherlands
- 15 primary care sites across Portugal, Porto, Portugal
- 15 primary care sites across Palma De Mallorca, Madrid, Murcia, Palma de Mallorca, Spain

IPD SHARING:
Plan to Share IPD: No